CLINICAL TRIAL: NCT06068257
Title: Translational Utility of Tumor-Derived FGF19 in a Novel Blood-Based Endocrine Suppression Approach
Brief Title: Tumor-Derived FGF19
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00005156
Record Dates: First submitted 2023-05-03; First posted 2023-10-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Breast Cancer; Healthy
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This study collects blood from breast cancer patients, colorectal patients, and healthy (no cancer) controls to identify biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Identify and test thresholds, specificity and sensitivity for a potential cancer associated biomarker protein, FGF19, (and associated markers) for detection in human blood in the blood of breast and colorectal in cancer patients, and see if occurs at higher rates than healthy controls

DETAILED DESCRIPTION:
This project seeks to develop and test a more convenient detection modality for colorectal cancer and to test feasibility for breast cancer screening through a blood based test for cancer detection. Because detection of cancer is a fundamental need to facilitate treatment and decrease patient mortality, the ultimate objective of this proposal is to test applicability and context for the blood test, especially for patients that either are not eligible or do not want to participate in currently approved screening protocols.

Colonoscopy and mammograms are gold standard cancer screening modalities that are recommended for detection of early-staged tumors, but there are many reasons why patients are noncompliant with participation in these screening modalities. Neither colorectal cancer nor breast cancer detection have reliable blood based cancer tests.

Availability of blood based cancer tests could increase patient compliance, as well as decrease the associated mortality in finding cancer at later stages. The Altomare laboratory has identified that FGF19 demonstrates unique characteristics that make it an attractive serum marker for this concept. This UCF research group has found that in studies using mice injected with human colorectal cancer cells, that FGF19 is secreted into blood by tumors. The findings support the concept that malignant FGF19 from certain tumors such as colorectal cancer can be leveraged in a diagnostic context to improve cancer detection and access to screening.

Both colorectal cancer and breast cancer patients are priority populations for the Florida Cancer Grant Programs. Importantly, FGF19 has not been tested for threshold, sensitive or specificity as a blood marker for colorectal cancer. Baseline FGF19 blood marker levels corresponding to colorectal cancer testing will be compared with those of another cancer type, breast cancer, where aberrant FGF19 levels have been implicated but also not tested. The investigators therefore also will test the applicability of serum FGF19 to detect breast cancer, which has dysregulation of FGF19 and its receptor in certain subtypes of breast tumors.

Objectives:

The primary marker that the investigators will look for is FGF19, a factor of normally restricted spatially to parts of the intestine and gall bladder, especially following a meal. The investigators will test in cancer patients whether FGF19 (or other associated markers) are higher in the blood of subset of cancer patients.

The investigators pose the question of whether FGF19 is actively secreted into blood by human tumors. In further examine its use as a blood biomarker, the investigators will address whether higher levels of FGF19 cutoffs can be detected in the blood of colorectal cancer or breast cancer patients over that of control participants. Successful completion of this goal will, for the first time, establish whether tumor production of FGF19 in human colorectal or breast tumors contributes to elevated levels in either, all or a subset of patients compared to blood levels in people without cancer.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll adult persons with breast cancer or colorectal cancer or no cancer (healthy controls) who are able to do a fasting blood draw.

(Pregnant women may choose to be in the study. The study procedures do not pose a risk to the safety of the unborn child or the woman.)

Exclusion Criteria:

* The study will not enroll persons who are unable or unwilling to provide informed consent.
* Adults unable to consent, individuals who are not yet adults, and prisoners will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants currently diagnosed with breast cancer and colorectal cancer, as well as, healthy participants who are currently cancer-free.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
To Identify and test thresholds, specificity and sensitivity for FGF19, (and associated markers) for detection in human blood of breast and colorectal in cancer patients, and see if occurs at higher rates than healthy controls. | 1 year
  The primary marker that the investigators will look for is FGF19, a factor of normally restricted spatially to parts of the intestine and gall bladder, especially following a meal. The investigators will test in cancer patients whether FGF19 (or other associated markers) are higher in the blood of subset of cancer patients.
  The investigator pose the question of whether FGF19 is actively secreted into blood by human tumors. In further examine its use as a blood biomarker, the investigators will address whether higher levels of FGF19 cutoffs can be detected in the blood of colorectal cancer or breast cancer patients over that of control participants. Successful completion of this goal will, for the first time, establish whether tumor production of FGF19 in human colorectal or breast tumors contributes to elevated levels in either, all or a subset of patients compared to blood levels in people without cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Altomare, PhD, Principal Investigator — University of Central Florida College of Medicine
Locations (1):
- Burnett School Biomedical Sciences, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided